CLINICAL TRIAL: NCT04045041
Title: A Guided Internet-based CBT Treatment for Provoked Vestibulodynia:a Randomized Controlled Trial
Brief Title: Internet-based Treatment for Provoked Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Monica Buhrman, PhD, licensed psychologist & psychotherapist, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180501
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Provoked Vestibulodynia; Vulvodynia, Generalized
Keywords: Provoked vestibulodynia; Exposure treatment; Cognitive behaviour therapy; Acceptance and commitment therapy; Pain; Internet-based; Vulvodynia
MeSH Terms: conditions — Vulvodynia; Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): 10 week internet-based acceptance and commitment therapy
  Interventions: Behavioral: Acceptance and commitment therapy
- Control group (No Intervention): Waiting-list control.

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — An acceptance based intervention with focus on exposure.
  Arms: Treatment group

SUMMARY:
Provoked vestibulodynia is a pain condition, which is associated with lower quality of life and discomfort. Furthermore, it is underdiagnosed and undertreated. Provoked vestibulodynia is defined as vulvar pain with no known cause. Provoked vestibulodynia can be generalized and involve several areas of the vulva. It can also be localized and involve only one area of the vulva. Pain is often provoked by touch or pressure but it can also be spontaneous or both. The life prevalence for vestibulodynia varies between 3-28 percent in different populations. Persons with vestibulodynia report more frequently anxiety-, depression- and stress- symptoms than the normal population.

The aim of the present study is to evaluate an internet-based treatment for vestibulodynia. The intervention will be based on Acceptance and commitment therapy (ACT) and cognitive behavior therapy with focus on exposure and acceptance.

DETAILED DESCRIPTION:
Patients suffering from vestibulodynia often experience psychological distress. Acceptance and commitment therapy (ACT) has been shown to be effective in treating psychological distress and pain. However delivering relevant treatment can be difficult due to logistics, cost and lack of personnel with required competence. Delivering ACT though the internet (iACT) is a novel approach, sidestepping logistical issues while lowering costs. There is however, a need to research this kind of treatment for persons with vestibulodynia.

This study will primarily investigate whether an ACT-treatment administered through the internet can be beneficial for patients suffering from provoked vestibulodynia. The treatment will be 10 weeks long. Participants will be randomized to the treatment program or a waiting-list control group. Analysis of possible mediating variables will be able to give insight into the internal workings of the treatment itself, further elucidating efficacy of specific interventions, data which will be useful in future developments of treatment design.

The treatment will consist of a 10-week period where participants would get access to a series of treatment modules, each addressing a separate problem area using ACT techniques. The treatment includes modules focuses on acceptance and exposure techniques. The participants will receive every week different exposure assignments. The platform used is an existing platform employed by the Pain Center at Uppsala university hospital for delivering internet based treatments.

The study will be conducted using a randomized controlled trial with a between-group design. Participants will be randomized to two groups, were one group will gain access to iACT treatment while the second group will be a wait-list control, and will gain access to the program once treatment of the active group is finished. A licensed psychologist will assess participants. In addition to online ACT modules, consisting of information, exercises and homework assignments, all participants will have regular contact by secure email-channel with a licensed psychologists or last-year psychology student under supervision. This contact will guide treatment, providing support, feedback on homework, and if necessary clarify treatment content and help with IT-related problems interfering with treatment adherence. After a year, participants will be invited to take part in a follow-up module, consisting of limited treatment recapitulation and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* suffer from provoked vestibulodynia/symptoms of vestibulodynia for three months or more or have been received the diagnosis vestibulodynia
* access to the internet
* 18 years old or older
* good knowledge of Swedish (since the material will be in Swedish)

Exclusion Criteria:

* suffer from serious psychological problems that requires clinical care or problems with addiction
* involved in an ongoing psychological treatment
* scheduled activity that will impede the participant to participate in the treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study was aimed at individuals with a vagina since it is a treatment for vestibulodynia.
Enrollment: 60 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Female sexual function index | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  It measures sexual dysfunction with 19 items. The answers are rated in a likert scale ranging from 0-5 regarding sexual activity. The results are presented in one total scale
Female sexual distress-scale | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  It measures distress related to sexual function with 13 items and an additional question. The answers are rated from Always, Often, Sometimes, Rarely and Never. The results are presented in one total scale

SECONDARY OUTCOMES:
Brunnsviken Brief Quality of Life Inventory (BBQ) | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  BBQ has a total of 12 items covering six life areas: Leisure, View on life, Creativity, Learning, Friends and Friendship, and View on self. All items are scored using the same response format, consisting of a five-step Likert rating scale, visually scored 0-4 with written anchor points at 0 (Strongly disagree) and 4 (Strongly agree). The BBQ total score is computed by summing the weighted satisfaction ratings, i.e. by multiplying the Satisfaction and Importance items for each life area and summing the six products for a total score (possible score range 0-96).
Pain severity scale in Multidimensional Pain Inventory (MPI) | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  The pain severity scale contains three items ranging from 0 to 6 (seven points) and measures pain intensity. The score is calculated by adding the score for each item divided by the number of items (scores range from 0-6). Higher scores indicate greater pain intensity.
Montgomery Åsberg Depression Rating Scale (MADRS-S) | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  The Montgomery Åsberg Depression Rating Scale measures depression symptom with 9 items.The respondents rate their symptoms on a scale that ranges from 0 to 6, where a higher value indicates a higher level of depressive symptoms. The score can range from 0-54, higher scores indicate more severe depressive symptoms e.g. a score >35 indicates a severe depression. The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
Generalised Anxiety Disorder 7-item scale (GAD-7) | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  Generalized Anxiety Disorder 7-item scale /GAD-7) measures anxiety with 7 items. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions. GAD-7 total score for the seven items ranges from 0 to 21.
Vaginal penetration cognition questionnaire (VPCQ) | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  The Vaginal penetration cognition questionnaire (VPCQ) measures cognitions regarding vaginal penetration are assessed where the participant score in a likert scale ranging from 0-6 in 22 statements. Possible answers range from "0 = not at all applicable" to "6 = very strongly applicable." The VPCQ consists of 5 subscales: Control Beliefs (4 items), Catastrophic and Pain Beliefs (5 items), Self-Image Beliefs (6 items), Positive Beliefs (5 items), and Genital Incompatibility Beliefs (2 items).
Chronic pain acceptance questionnaire (CPAQ) | Baseline-, mid-(week 5), post-(at 10 weeks) and follow up- measure (6months)
  Chronic pain acceptance questionnaire (CPAQ) measures with 20 items acceptance related to pain and an aspect of psychological flexibility. It is a process variable and consists of two subscales, Willingness and Engagement. Items are rated on a scale from 0 (never true) to 6 (always true).Higher scores denote greater activity engagement and pain willingness.The total score is also reported, higher scores is associated with higher levels of acceptance.
Committed Action Questionnaire-8 (CAQ-8) | Baseline-, mid-(week 5), post-(at 10 weeks) and follow up- measure (6months)
  Committed Action Questionnaire (CAQ-8) measures commitment, an aspect of psychological flexibility. It is a process variable and consists of 8 items. lease rate the truth of each statement as it applies to you by circling a number. The rating scale ranges from 0(never true)to 6 (always true). The total score represents an individual's general propensity to persist in goal-directed behaviour, capturing both positive and negative aspects of the construct. Higher values indicating higher levels of committed action.
Mindful Attention Awareness Scale (MAAS) | Baseline-, mid-(week 5), post-(at 10 weeks) and follow up- measure (6months)
  The Mindful Attention Awareness Scale (MAAS) is a 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present. Mindful attention awareness, an aspect of psychological flexibility. It is a process variable. The responder mark their response in a 1-6 scale and indicate how frequently or infrequently the person currently have each experience. To score the scale, the mean of the 15 items is calculated. Higher scores reflect higher levels of dispositional mindfulness.
Treatment credibility scale (TCS) | After the first treatment week
  The treatment credibility scale (TCS) measures how credible the treatment is perceived by the participant where the participant rates five statements. Every item i rated on a scale from 1 to 10, the last question is rated from 0% to 100%. The score is calculated by adding the score for each item.Higher values are associated with higher expectancy and credibility.
CHAMP Sexual Pain Coping Scale (CSPCS), | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  Sexual Pain Coping Scale (CSPCS) measure avoidance and endurance coping behaviors during penetration with 12-item. This measure consists of three sub-scales: avoidance, endurance and alternative strategies. Respondents rate their agreement of each statement between 1 ("Never true") and 7 ("Always true"). Total scores range from 4-28 on each sub-scale.12 items that measures cognitions and emotions related to sex and sexual pain
Quality of dyadic relationship (QDR-36) | Baseline-, post-(at 10 weeks) and follow up- measure (6months)
  Measures 5 dimensions (Dyadic Consensus, Dyadic Satisfaction, Dyadic Sensuality, Dyadic Cohesion and Dyadic Sexuality)of a relationship with 36 items. Answers are rated in a scale that ranges from 1-6, an average score is calculated for every dimension. The average in every dimension is summed and an index is calculated which ranges from 5-30. The quota for the total questionnaire ranges from 6 to 1. Higher scores indicate good perceived quality in the relationship while lower scores indicate lower quality in the relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Buhrman, PhD, Principal Investigator — Uppsala University; Lance McCracken, Professor, Study Chair — Uppsala University
Locations (1):
- Department of psycholology, Uppsala university, Uppsala, Uppland, Sweden